CLINICAL TRIAL: NCT05388591
Title: Evaluation of Musicotherapy (Application Music Care) on Pain During Wound Closure in the Emergency Department : a Randomized Controlled Trial.
Brief Title: Evaluation of Musicotherapy on Pain During Wound Closure in the Emergency Department
Acronym: EMERGENCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022/CHU/10
Record Dates: First submitted 2022-05-19; First posted 2022-05-24 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: Wounds Injuries
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Musicotherapy (Experimental)
  Interventions: Other: Musicotherapy
- Standard care (No Intervention)

INTERVENTIONS:
Other: Musicotherapy — Music listening with the application Music Care (style of music chosen by the patient) during wound suturing
  Arms: Musicotherapy

SUMMARY:
To evaluate the effectiveness of music listening (with a musicotherapy application Music Care) on patients pain associated with care during wound suturing in the Adults emergency unit.

DETAILED DESCRIPTION:
BACKGROUND - Music therapy is known as an effective adjuvant treatment for the management of physical pain and anxiety. It is recognised in various medical fields. Wound suturing in the Emergency Department is a potentially stressful and painful experience for patients.

OBJECTIVE - To evaluate the effectiveness of music listening (with a musicotherapy application Music Care) on patients pain associated with care during wound suturing in the Adults emergency department.

METHODS - Therefore, a prospective, randomised, open-label, multi-centre interventional will be conducted in two Adults Emergency departments of the Reunion Island University hospitals.

Patients over 18 years old admitted to the Adults Emergency Departments with a suturable wound (at least one stitch), able to understand and express themselves will be included.

The primary outcome is the comparison of maximal VAS score between the two groups. Secondary outcomes are the absolute change in heart rate, systolic and diastolic blood pressure, respiratory rate, absolute change in anxiety score, suture duration related to the number of stitch, overall patient and practitioner satisfaction.

The baseline data collection includes patient age and sex, pain and stress VAS and biological parameters (heart rate, blood pressure, respiratory rate) at admission in box and immediately after suturing.

In order to demonstrate a difference of 10mm on VAS with a standard deviation of 20mm, a power of 90% and an alpha risk of 0,05, the number of subjects required is 192.

A multivariate analysis was performed on the association between exposure : music/no music and the judgement criteria. Subgroup analyses are planned for age, gender, additional analgesia used, location, duration of analgesia used, location, duration of suture and number of stitches.

EXPECTED RESULTS - Thanks to music therapy, a decrease of pain and anxiety associated with sutures in the Emergency room is expected, but also an improvement in the working conditions hospital physicians in the emergency room.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years admitted to ER with suturable wound (at least 1 stitch)
* able to understand and express oneself
* giving free, informed and written consent signed by the participant and the investigator

Exclusion Criteria:

* who has a severe wound with suspected open fracture or requiring surgical exploration in the operating room
* with severe hearing loss or deafness, speech disorders or any acute or chronic condition that compromises listening (at the investigator's discretion), musicogene epilepsy
* no social security cover
* unable to decide for himself or herself (at the discretion of the investigator): confused patient, foreign language not understood by the investigator, severe acute intoxication, patient with severe neurological or psychiatric comorbidity
* under judicial protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2022-06-14 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
Evaluate the efficacy of musicotherapy on maximal pain associated with wound injury closure in emergency unit | Day 1
  Comparison of maximal pain using visual analogic scale score between the two groups (scale ranking from 0 to 10, with 0 meaning better score (no pain/no anxiety) and 10 the worse score (maximal pain/anxiety).

CONTACTS AND LOCATIONS:
Overall Officials: Thien-Kim DINH, MD, Principal Investigator — CHU La Réunion
Locations (2):
- Reunion (2):
  - CHU de la Réunion, Saint-Denis
  - CHU de la Réunion, Saint-Pierre

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Charron M, Daniel M, Guihard B, Gokalsing E, Faure L, Bruneau L, Dinh K. Evaluation of a web app-based music intervention on pain during wound closure in the emergency department: The EMERGENCE randomized controlled trial. Anaesth Crit Care Pain Med. 2025 Aug;44(4):101545. doi: 10.1016/j.accpm.2025.101545. Epub 2025 May 21. PMID 40409580